CLINICAL TRIAL: NCT05912153
Title: SPECT-CT Versus MRI for the Diagnosis of Symptomatic Osteoarthritis in the Ankle, Hind- and Midfoot.
Brief Title: SPECT-CT Vs MRI for the Diagnosis of Osteoarthritis in the Foot and Ankle
Status: Recruiting | Type: Observational
Sponsor: Martini Hospital Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: ProSPECT study
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-05

CONDITIONS: Osteoarthritis Ankle; Osteoarthritis
Keywords: SPECT/CT; MRI; osteoarthritis; Foot and/or Ankle
MeSH Terms: conditions — Osteoarthritis | interventions — Single Photon Emission Computed Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: SPECT/CT — SPECT/CT of the foot and ankle
Diagnostic Test: MRI — MRI of the foot and ankle

SUMMARY:
The diagnose of symptomatic osteoarthritis in the ankle, mid- and hind foot remains challenging. There is no gold standard for the work-up and various hospitals use different protocols. Current literature shows a promising role for SPECT-CT imaging in ankle, hind- and midfoot OA. In a previous study investigating the role of SPECT-CT in a reproducible group we have observed a change in diagnosis in 53% when SPECT-CT data was added to the data of conventional workup alone. In 26% of patients addition of SPECT-CT data resulted in change of the original treatment plan. To our knowledge no prospective studies are available on this subject for both SPECT-CT and MRI. In our clinic both SPECT-CT and MRI are used in the work-up for patients with ankle, hind- and midfoot pain. Although we experience good result with SPECT-CT, MRI might be able to detect symptomatic OA as well. Moreover MRI provide more information about soft tissue and is less harmful for the patient in comparison to SPECT-CT. The aim of this study is to determine the diagnostic performance of SPECT-CT and MRI when used routinely in patients with symptomatic OA of the ankle, hind- and midfoot.

DETAILED DESCRIPTION:
Objective: The objective is to determine diagnostic performance of SPECT-CT and MRI when used routinely in patients with symptomatic OA of the ankle, hind- and midfoot.

Study design: Prospective cohort study.

Study population: All patients ≥18years old, referred to the Martini Hospital Groningen department of Orthopedic surgery with suspected symptomatic osteoarthritis of the foot and ankle and rest pain of NRS ≥4.

Main study parameters/endpoints: Main parameters will be the diagnostic performance (a.o. sensitivity and specificity, positive and negative predictive value)of SPECT-CT and MRI.

The standard work up consist of questionnaires, detailed physical examination, conventional radiographic, MRI, SPECT-CT imaging and ultrasound guided injections. There are no additional risks for participating in this study compared to current standardised hospital workup.

ELIGIBILITY:
Inclusion Criteria:

* Suspected symptomatic ankle, hind- or midfoot OA
* Informed consent
* Age ≥ 18 years
* Average NRS ≥4 over the past week.

Exclusion Criteria:

* Contraindication for surgery
* Contraindication for SPECT-CT or MRI
* Contraindication for intra-articular injections
* Isolated forefoot pathology
* Fracture, ligamentous or tendon injury of the ankle, hind- and/or midfoot trauma within one year before presentation
* History of neurological disease
* History of foot and/or ankle surgery (affected side)
* Inability to read and understand the written information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients subjects will be all patients referred to the Martini Hospital Groningen with suspected OA of the foot and ankle meeting our inclusion criteria. In total 369 patients will be included. A sample of two months showed that 68 new eligible patients were presented at the outpatient clinic with a prevelence of OA in 85%. We assume that at least 50% of the eligible patients are willing to participate in this study, so it is expected that within 24-30 months all patients can be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of SPECT/CT and MRI | 1 year
  Primary objective is to determine overall diagnostic performance (in terms of sensitivity + specificity, positive and negative predictive values, positive and negative likelihood ratios, and diagnostic odds ratio) of SPECT-CT and MRI for diagnosing symptomatic OA in the ankle, hind- and midfoot.

CONTACTS AND LOCATIONS:
Overall Officials: Tom van Raaij, MD/PhD, Principal Investigator — Martini Ziekenhuis
Locations (1):
- Martini Hospital, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Only deidentified data will be available upon reasonable written request in conjunction with appropriate data use agreement.